CLINICAL TRIAL: NCT03592849
Title: The Efficacy and Safety of Collagen Scaffold Loaded With Umbilical Cord Derived Mesenchymal Stem Cells in Infertile Women With Thin Endometrium or Endometrial Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yali Hu, Professor，Chief Physician of Obstetrics and Gynecology, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC201700101
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Infertility, Female; Endometrium
Keywords: thin endometrium; infertility
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UC-MSCs therapy (Experimental): transplant collagen scaffold loaded with UC-MSCs to treat infertility caused by thin endometrium or endometrial scarring
  Interventions: Procedure: UC-MSCs therapy

INTERVENTIONS:
Procedure: UC-MSCs therapy — After history taking, physical examination, ultrasound examination and hysteroscopy examination，infertile women diagnosed with thin endometrium or endometrial scarring will be included in the clinical trial. A collagen scaffold loaded with UC-MSCs will be transplanted into the uterine cavity during hysteroscopy, and participants will receive hormone replacement therapy before and after the treatment. Postoperative observations including ultrasound examination once a month for 3 times and hysteroscopy in the third month after first UC-MSCs therapy. Those whose endometrium is suitable for pregnancy will be recommended attempting conception actively. The next round of cell therapy will be conducted 3 cycles after the first month if the endometrial growth is unsatisfactory.
  Other Names: collagen scaffold

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the collagen scaffold loaded with umbilical cord derived mesenchymal stem cells (UC-MSCs) in infetile women with thin endometrium or endometrial scarring.

ELIGIBILITY:
Inclusion Criteria:

1. Infertile patients with clear fertility desires
2. Diagnosed with thin endometrium or endometrial scarring for whom drugs and surgical interventions were ineffective
3. 20-42 years old
4. Normal ovarian function or with frozen embryos
5. Willing to actively cooperate with postoperative follow-up

Exclusion Criteria:

1. With abnormal chromosome karyotype
2. With other uterine diseases including large intramural myomas, severe endometriosis, severe adenomyosis, severe congenital uterine malformations, endometrial tuberculosis, vaginitis and endometritis
3. Systemic diseases: hypertension, diabetes, and so on
4. Contraindications to pregnancy
5. Contraindications to hormone replacement therapy
6. Medical history of pelvic tumors or receiving pelvic radiotherapy
7. Involved in other clinical studies
8. Unable to adhere to the follow-up

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 20 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
endometrial thickness | 12 months
  endometrium thickness evaluated by transvaginal sonography during late proliferating phase

SECONDARY OUTCOMES:
ongoing pregnancy rate | 24 months
  the presence of a living intrauterine fetus on TVU at the 12th week of gestation
live birth rate | 24 months
  a live born baby ≥28 weeks of gestation
endometrial blood flow | 6 months
  uterine blood flow evaluated by transvaginal sonography

OTHER OUTCOMES:
menstrual blood volume | baseline and 6 month postoperation
  the change of menstrual blood volume after surgery compared with pre-operation
adverse event rate | 30 months
  the occurrence of infections、allergies、abdominal pain postoperation

CONTACTS AND LOCATIONS:
Overall Officials: Yali Hu, MD,PhD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Within six months after the trial complete